CLINICAL TRIAL: NCT03309163
Title: Effect of Tramadol in Prevention of Postpartum Depression
Acronym: ETPPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Hong Li, Director, Department of Anesthesiology, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ETPPD Trail
Record Dates: First submitted 2017-09-28; First posted 2017-10-13 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Caesarean Section
MeSH Terms: interventions — Tramadol; Hydromorphone; Ropivacaine; Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group T (Active Comparator): All patients receive the patient-controlled intravenous analgesia with Tramadol.
  Interventions: Drug: Tramadol
- Group H (Placebo Comparator): All patients receive the patient-controlled intravenous analgesia with Hydromorphone.
  Interventions: Drug: Hydromorphone
- Group E (Placebo Comparator): All patients receive the patient-controlled epidural analgesia with Ropivacaine.
  Interventions: Drug: Ropivacaine (Epidural analgesia)

INTERVENTIONS:
Drug: Tramadol — Patient-controlled intravenous analgesia with Tramadol
  Arms: Group T
Drug: Hydromorphone — Patient-controlled intravenous analgesia with Hydromorphone
  Arms: Group H
Drug: Ropivacaine (Epidural analgesia) — Patient-controlled epidural analgesia with Ropivacaine.
  Arms: Group E

SUMMARY:
The incidence of postpartum depression in Europe and the United States is about 10%, while in China the incidence rate of 15.7-39.8%. Postpartum depression is one of the most common diseases of perinatal distress, but the current research of high-quality prevention and treatment of postpartum depression is still very lack. The study suggests that the risk of postpartum depression in cesarean delivery is significantly higher than that in vaginal delivery. Therefore, postpartum depression in cesarean delivery may require more attention and treatment.Tramadol is a non-opioid central analgesic that relieves common to severe pain, and tramadol has an inhibitory effect on norepinephrine and serotonin systems and has the potential to reduce depression and anxiety. Therefore, for the analgesic demand and antidepressant demand for maternal who undergoing cesarean section, tramadol may be an optimized and effective analgesic for the prevention and treatment of postpartum depression.

DETAILED DESCRIPTION:
This study was designed according to a prospective, randomized, controlled clinical trial. Randomized subjects were randomly assigned to different analgesic drug-treated groups according to the random number induced by SPSS software. All three analgesic treatments were routinely used for clinical analgesia; Anesthesia, surgery, postoperative treatment are in accordance with clinical practice. The investigators conducted a postoperative questionnaire survey and psychological diagnosis for all patients. And blood sample was collected from patients before and 48 hours after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* 20 years old ≤ age ≤ 40 years old;
* ASA score I-Ⅱ;
* uncomplicated and singleton full-term pregnancy;
* voluntarily to receive cesarean section and postoperative controlled analgesia;
* consent to participate the study.

Exclusion Criteria:

* with history of mental disorders or psychotropic substances use;
* with history of neurological diseases such as epilepsy
* with history of previously known diagnosed depression;
* with suicidal ideation or history of suicide;
* with history of drug，alcohol or opioid abuse;
* with monoamine oxidase (MAO) inhibitor treatment at present or in the past 14 days;
* participating in other clinical studies
* with severe heart disease, brain disease, liver disease and kidney disease;
* be allergic to tramadol or opioids;
* with any contraindication for combined spinal epidural anesthesia;
* incapable of communication or cooperation.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1230 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
The incidence of postpartum depression | At 4 weeks after the surgery
  Diagnosed according to DSM-5 diagnostic criteria for postnatal depression

SECONDARY OUTCOMES:
The incidence of postpartum depression | At 3 months after the surgery
  Diagnosed according to DSM-5 diagnostic criteria for postnatal depression
EPDS scores | At 4 weeks and 3 months after the surgery
  Measured using Edinburgh Postnatal Depression Scale
GAD-7 scores | At 4 weeks and 3 months after the surgery
  Measured using Generalized Anxiety Disorder Scale
QoR-15 scores | 48 hours after the surgery
  Measured using Quality of recovery 15
Pain intensity | At 6, 12, 24 and 48 hours after the surgery
  Pain VAS at 6, 12, 24 and 48 hours after the surgery
Norepinephrine and serotonin levels in the blood | At 48 hours after the surgery
  Norepinephrine and serotonin concentration in the blood at 48 hours after the surgery

OTHER OUTCOMES:
Early walking time | During hospitalization, an average of 36 hours
  The time for patient to independently activity
Hospital stays | During hospitalization, an average of 72 hours
  The time for patient to stay in hospital after the surgery
Pain intensity | At 3 months after the surgery
  Postoperative pain intensity that evaluated by questionnaire at 3 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hong Li, M.D., Principal Investigator — Department of Anesthesiology, Xinqiao Hospital, Third Military Medical University
Locations (1):
- Xinqiao Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu Z, Zhao P, Peng J, Fang L, Ding J, Yan G, Wang Y, Zhu J, Wang D, Li Y, Chen Z, Zhang Q, Deng Q, Duan G, Zuo Z, Li H. A Patient-Controlled Intravenous Analgesia With Tramadol Ameliorates Postpartum Depression in High-Risk Woman After Cesarean Section: A Randomized Controlled Trial. Front Med (Lausanne). 2021 May 27;8:679159. doi: 10.3389/fmed.2021.679159. eCollection 2021. PMID 34124111
- [Derived] Duan G, Wu Z, Zhao P, Peng J, Chen Z, Zhang Q, Xu R, Li H. Protocol for a randomised, double-blind, placebo-controlled trial to explore the effect of tramadol in the prevention of postpartum depression (ETPPD). BMJ Open. 2018 Oct 21;8(10):e022538. doi: 10.1136/bmjopen-2018-022538. PMID 30344172